CLINICAL TRIAL: NCT01999907
Title: Vitamin D vs. Placebo in the Prevention of Viral-induced Exacerbations in Preschoolers With Asthma: a Pilot RCT
Brief Title: Vitamin D to Reduce Colds and Asthma Attacks in Young Children
Acronym: DIVA-pilot
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Professor Francine Ducharme, Professor & Pediatrician, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VD0001; 12140 (Other Grant/Funding Number: Thrasher Research Fund)
Record Dates: First submitted 2013-11-25; First posted 2013-12-03 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: Asthma
Keywords: asthma; virus diseases; pediatric; RCT; steroid
MeSH Terms: conditions — Asthma; Virus Diseases | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): bolus placebo given in a 2ml dose by mouth at baseline. This group receives daily vitamin D supplement by mouth for the 6 month study (400IU cholecalciferol per day).
  Interventions: Dietary Supplement: daily vitamin D supplement; Other: Placebo
- Vitamin D (Active Comparator): Vitamin D (100,000IU) bolus in a 2ml dose by mouth given at baseline. This group receives a daily vitamin D supplement by mouth for 6 months (400IU cholecalciferol per day).
  Interventions: Dietary Supplement: Vitamin D; Dietary Supplement: daily vitamin D supplement

INTERVENTIONS:
Dietary Supplement: Vitamin D — 100,000IU cholecalciferol given in a 2ml dose by mouth at baseline.
  Other Names: cholecalciferol
  Arms: Vitamin D
Dietary Supplement: daily vitamin D supplement — Each group receives a daily vitamin D supplement for 6 months, providing 400IU per day.
  Other Names: cholecalciferol (Pediavit)
Other: Placebo — placebo given in a 2ml dose by mouth at baseline.
  Arms: Placebo

SUMMARY:
Viral infections are the main cause of asthma attacks in preschoolers, an age group with the highest rate of emergency visits due to asthma. While high doses of inhaled or oral corticosteroids provide benefits, these have been associated with adverse outcomes. Most asthmatic children have lower blood levels of vitamin D compared to non-asthmatic children. Low vitamin D level has been linked to more frequent and more severe asthma attacks as well as with higher dose requirement of inhaled corticosteroid. Recent studies show that vitamin D supplements can reduce the number of asthma attacks triggered by viral infections in children. Unfortunately, most people forget to take vitamin D every day during the fall and winter season as recommended in Canada. A solution is to give a vitamin D bolus by mouth. This has been shown to safely and effectively increase vitamin D levels in children. The investigators hypothesise that a vitamin D bolus given in clinic will sufficiently increase the blood level of vitamin D to prevent the expected winter decline in vitamin D, compared with placebo in preschool-aged children with asthma. This six-month pilot randomized controlled trial aims to: (1) show that a vitamin D bolus is superior to placebo in raising vitamin D levels; (2) record the number of asthma attacks and viral infections in enrolled participants; and (3) identify problems that may call for protocol changes.

ELIGIBILITY:
Inclusion Criteria:

* children aged 1-5 years
* physician-diagnosed asthma as per GINA guidelines
* upper respiratory tract infections as the main asthma exacerbation trigger
* ≥4 respiratory infections in the past 12 months
* ≥1 exacerbation requiring rescue oral steroids in the past 6 months or ≥2 in the previous 12 months.

Exclusion Criteria:

* extreme prematurity (<28 weeks gestation)
* infants <12 months of age
* breastfed infants with no vitamin D supplementation
* recent (<1 year) immigrants from countries where rickets and malnutrition prevalent
* other chronic respiratory disease (broncho-pulmonary dysplasia; cystic fibrosis)
* endocrine disorder of calcium/ vitamin D metabolism
* disorder/ disease with associated malabsorption (inflammatory bowel disease)
* kidney/ liver disease
* sickle cell anemia
* medications known to interfere with bone metabolism/ vitamin D levels
* vitamin D supplementation >1000 IU/ day in past 3 months
* unable to attend medical visit in 3-4 months
* plan to leave the province during the next 6 months.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2013-11; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
serum Vitamin D | 3 months
  mean change in serum vitamin D from baseline to 3 months

SECONDARY OUTCOMES:
adequate serum vitamin D | 3 months
  difference in the proportion of children with serum vitamin D ≥75nmol/L at 3 months

OTHER OUTCOMES:
exacerbations requiring oral corticosteroids | 6 months
  number of patients with one or more exacerbations requiring oral steroids, as documented by pharmacy dispensation records and medical records
number of viral infections | 6 months
  number of patients/person-month of observation documented two days
  1. parent-reported on the Canadian Acute Respiratory Illness and Flu Scale and
  2. Positive viral presence, determined by polymerase chain reaction on nasal sample
Hypercalciuria | any point during the 6 months
  urinary calcium: creatinine ratio >1.25 (1-2 years) and >1 (2-5 years) mmol/mmol
Cytokine/ chemokine profile | 10 days
  change in serum cytokine/ chemokine profile from baseline to 10 days post-bolus dose
duration of viral infections | in the event of a cold during the 6 months
  number of days with respiratory tract symptoms as reported on the parent completed Canadian Acute Respiratory Illness & Flu Scale
severity of exacerbations | in the event of an exacberbation during the 6 months
  1. area under the curve for β-agonist use as documented by parent of the 'Asthma Flare-Up Diary for Young Children';
  2. need for hospital admission
duration of exacerbations | in the event of an exacerbation during the 6 months
  Number of days with asthma symptoms as reported on the parent-reported 'Asthma Flare-Up Diary for Young Children'
participant retention | 6 months
  percentage of patients retained until 6 months after randomization
protocol adherence | 6 months
  1. participant attendance to all 4 home and clinic visits
  2. percentage of patients with all 4 blood and urine tests collected
  3. percentage of analyzable viral nasal swabs returned.

CONTACTS AND LOCATIONS:
Overall Officials: Francine M Ducharme, Principal Investigator — St. Justine's Hospital
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Huey SL, Acharya N, Silver A, Sheni R, Yu EA, Pena-Rosas JP, Mehta S. Effects of oral vitamin D supplementation on linear growth and other health outcomes among children under five years of age. Cochrane Database Syst Rev. 2020 Dec 8;12(12):CD012875. doi: 10.1002/14651858.CD012875.pub2. PMID 33305842
- [Derived] Jensen ME, Mailhot G, Alos N, Rousseau E, White JH, Khamessan A, Ducharme FM. Vitamin D intervention in preschoolers with viral-induced asthma (DIVA): a pilot randomised controlled trial. Trials. 2016 Jul 26;17(1):353. doi: 10.1186/s13063-016-1483-1. PMID 27456232